CLINICAL TRIAL: NCT01556074
Title: Evaluation of Yoga for Sleep Disturbances in Insomnia and Posttraumatic Stress Disorder
Brief Title: Evaluation of Yoga for Sleep Disturbances in Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Sat Bir Khalsa, PhD, Assistant Professor in Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000263; F32AT006092-01A1 (NIH); 18180 (Other Grant/Funding Number: BBRF)
Record Dates: First submitted 2012-03-08; First posted 2012-03-16 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Post Traumatic Stress Disorder; Insomnia
Keywords: Post traumatic stress disorder; PTSD; Insomnia; Sleep; Yoga; Meditation; Mental Health; Sleep Quality; Actigraphy; Sleep Diaries; Autonomic; Social Health; Interoception; Attention Regulation; Emotion Regulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yoga treatment (Experimental)
  Interventions: Behavioral: Yoga treatment

INTERVENTIONS:
Behavioral: Yoga treatment — Biweekly 90-minute group yoga classes for 8 weeks and on non-class days participants will be asked to devote 15 minutes per day to a prescribed home yoga practice.

SUMMARY:
The primary objective of this preliminary study is to estimate sleep outcome effect sizes and determine feasibility for a novel yoga treatment of insomnia in participants with post traumatic stress disorder (PTSD). Additional objectives are to evaluate relationships of sleep outcomes with measures of other PTSD symptoms, psychosocial health and possible mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female adults at least 18 years of age.
* A DSM-IV-TR diagnosis of post-traumatic stress disorder (PTSD).
* Naïve to yoga and other meditative practices, defined as less than one hour per week for the past 6 months.
* Potential subjects receiving ongoing medical or psychological treatment are eligible, as long as treatment remains stable over the course of the study and does not include more than one hour weekly of mind-body medicine (strategies directly related to meditation and yoga).
* No more than 2 alcoholic or caffeinated drinks/day
* No illicit drug use
* Potential subjects are eligible if they have been on stable dosage (not PRN) of medication for PTSD symptoms including sleep disturbances and any medication that may influence sleep for at least 6 weeks prior to the study, and be willing to continue with same dosage for the duration of the study.
* No current substance abuse, defined as diagnosis of substance abuse or dependence disorder within the past year, and/or in/outpatient treatment for substance abuse or dependence in the past 6 weeks.
* No transcontinental travel over the course of the study.
* No night-shift or rotating shift work over the course of the study.
* Insomnia based on the American Academy of Sleep Medicine's Research Diagnostic Criteria (RDC) for insomnia due to a mental health disorder
* Potential subjects are eligible to participate in this study if they have sufficient mental and physical ability to fully participate in the parameters of the study. Subjects must be able to understand and comply with instructions in the group yoga sessions and home practice, complete questionnaires, participate in clinical interviews, and take part in all data collection activities. Subjects with severe mental or physical concerns that may prevent them from understanding and/or complying with the treatment will be excluded. For example, potential subjects confined to wheelchairs will not be eligible, although subjects with artificial limbs who are able to reasonably participate in the intervention may be deemed eligible. These determinations will be made during discussions with potential subjects on a case by case basis during the screening process.

Exclusion Criteria:

- Potential subjects are ineligible if pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality measured by wrist actigraphy and daily sleep diaries | Averages of: 2-week pre-treatment baseline; last 2 weeks of treatment; 2-week long-term follow-up occuring 3-months post-treatment

SECONDARY OUTCOMES:
Acceptability of yoga program as measured by a 2-item Yoga Evaluation Form (End) and a 2-item Yoga Evaluation Form (Followup) | One occurrence at 1 week following intervention, one occurrence at 3 months post-intervention
Treatment adherence as measured by attendance to group yoga classes and play count monitoring of mp3's for home practice on non-class days | Averages over duration of intervention (8 weeks total)
Accrual rate calculated from recruitment and consent information | Monthly for duration of recruitment period (expected to be 3 months per cohort, up to 6 to 9 months for 2 to 3 cohorts total)
Attrition rate calculated from disempanelment information | Monthly for duration of data collection and treatment (approximately 6 months per cohort, up to 18 months for 2 to 3 cohorts total)
Change in PTSD symptoms as measured by the 17-item, self-reported PTSD Checklist-- Civilian version (PCL-C) | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in 10-min segment of a seated 30-min electrocardiogram (ECG) recording | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in emotional distress as measured by short forms of the Patient Reported Outcomes Measurement System (PROMIS) instruments for anxiety (4 items), depression (4 items) and anger (8 items) | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in social health as measured by short forms of the Patient Reported Outcomes Measurement System (PROMIS) instruments for social functioning (4 items), social functioning satisfaction (4 items) and social isolation (6 items) | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in interoception as measured by the 32-item self-reported Multidimensional Assessment of Interoceptive Awareness scale (MAIA) | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in emotion regulation as measured by the Difficulties in Emotion Regulation Scale (DERS) | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention
Change in sleep disturbance and sleep-related impairment as measured by two PROMIS scales | Once at 1-week before intervention, once at 1 week post-intervention, once at 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Noggle Taylor, PhD, Principal Investigator — Emory University; Sat Bir S Khalsa, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States